CLINICAL TRIAL: NCT03363048
Title: Effects of Subsidies and Prohibitions on Household Nutrition in a Food Benefit Program
Brief Title: Grocery Assistance Program Study for Families
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00002037
Record Dates: First submitted 2017-11-29; First posted 2017-12-05 (Actual); Last update posted 2020-11-10 (Actual); Status verified 2020-11

CONDITIONS: Nutritional Quality; Food Insecurity; Food Legislation; Healthy Diet; Food Stamp Program
Keywords: Food restrictions/incentives; Food Stamp program; Policy change; Supplemental Nutrition Assistance Program (SNAP)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Restricted (Experimental)
  Interventions: Behavioral: Restricted
- Restriction plus Incentive (Experimental)
  Interventions: Behavioral: Restriction plus Incentive
- Control (No Intervention)

INTERVENTIONS:
Behavioral: Restricted — Certain foods and beverages are not allowed to be purchased with food benefit dollars.
  Arms: Restricted
Behavioral: Restriction plus Incentive — Certain foods and beverages are not allowed to be purchased with food benefit dollars; 30% of the total dollars spent toward the purchase of certain foods result are added to their food benefit dollars.
  Arms: Restriction plus Incentive

SUMMARY:
An experimental trial will be conducted whereby a Supplemental Nutrition Assistance Program (SNAP)-like food benefit program will be implemented in 240 SNAP eligible households. Baseline and follow up measures will include three 24-hour dietary recalls; household food purchase receipt collection; and household food security questions. The individual level measures will be collected from the adult most responsible for food shopping and a child in the household. After baseline measures are completed households will be randomized to one of three conditions: 1) restriction (not allowed to buy sugar sweetened beverages, sweet baked goods, or candies with food benefits); 2) restriction paired with an incentive (30% financial incentive on fruits and vegetables and restriction of purchase of sugar sweetened beverages, sweet baked goods, or candy with food benefits); or 3) control (no incentive or restrictions). Households in all conditions will be given a debit card that will have funds added monthly for a five month period. The dollar amount placed on the card monthly will be similar to the amount the household would receive if enrolled in SNAP. All participants will be instructed to use the debit card for food purchases only, and they'll be told they shouldn't use the card to purchase items currently non-eligible for purchase with SNAP benefits (e.g. alcohol, food from restaurants). Those in the restriction condition will also be told they cannot use the card to buy sugar sweetened beverages, sweet baked goods, or candies. They may purchase these foods using their own money, but not the debit card. Those in the restriction plus incentive condition will receive the instructions provided to the restriction group plus they will be told that they'll receive a 30% bonus for fruits and vegetables purchased using their debit card. Analyses will determine whether the nutritional quality of the diet at follow-up differs between experimental groups.

ELIGIBILITY:
Inclusion Criteria:

* SNAP-eligible household
* at least one child between the ages of 3-11
* Less than or equal to 6 people in the household
* Primary food shopper
* Ability and willingness to collect and submit household food purchase receipts for 22 weeks
* Willingness to attend two study visits
* willingness to complete three dietary recalls at both baseline and follow-up
* not planning to apply for SNAP in the next 5 months
* ability to speak and understand either Spanish or English

Exclusion Criteria:

* households that are not SNAP-eligible
* no children in household between the ages of 3-11
* not primary food shopper
* 7 or more people in household
* inability to collect and submit household food purchase receipts for 22 weeks
* unwillingness to comply with study measures
* inability to speak or understand Spanish or English
* planning on applying for SNAP within the next 5 months.

Min Age: 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 646 (Actual)
Dates: Start 2018-05-02 (Actual); Primary Completion 2019-10-06 (Actual); Study Completion 2019-10-06 (Actual)

PRIMARY OUTCOMES:
Overall Nutritional Quality as measured by the Healthy Eating Index (HEI)-2015 score | 18 weeks
  Overall Nutritional Quality obtained from average intake of three dietary recalls at both baseline and follow-up.

SECONDARY OUTCOMES:
Total Energy Intake | 18 weeks
Scores of 3 components (whole fruits, total vegetable, and added sugar) of the HEI-2015 | 18 weeks
Household food insecurity | 18 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- University of Minnesota, School of Public Health, Division of Epidemiology & Community Health, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be placed on the Open Science Framework in compliance with Laura and John Arnold Foundation (LJAF) policies.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Data will be made available upon publication of the primary outcomes manuscript and will be posted indefinitely.
URL: https://osf.io/